CLINICAL TRIAL: NCT00108329
Title: 5449 Genetics, Weight Loss and Glucose Metabolism in Older Obese Men
Brief Title: Weight Loss in Diabetic, Older Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AGCG-005-00F
Record Dates: First submitted 2005-04-14; First posted 2005-04-15 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2007-04

CONDITIONS: Metabolic Syndrome X
Keywords: aging; exercise; metabolic syndrome; insulin resistance
MeSH Terms: conditions — Metabolic Syndrome; Motor Activity; Insulin Resistance

INTERVENTIONS:
Behavioral: Weight Loss

SUMMARY:
This study examines the effects of weight loss and aerobic exercise training on sugar metabolism and other risk factors for heart disease in obese older individuals.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years,
* Body mass index (BMI) > 27kg/m(2),
* No prior history of diabetes or coronary disease,
* Sedentary

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2003-04; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Locations (1):
- VA Maryland Health Care System, Baltimore, Maryland, United States